CLINICAL TRIAL: NCT05742516
Title: Does Galactooligosaccharide Supplementation Enhance Nutrient Availability in Physically Active Individuals
Brief Title: Does Galactooligosaccharide Enhance Nutrient Availability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Clasado Biosciences (Unknown)
Responsible Party: Principal Investigator, Adam Collins, Postgraduate Research Student, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 8779
Record Dates: First submitted 2023-02-02; First posted 2023-02-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Exogenous Carbohydrate Oxidation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOS (Experimental): Galactooligosaccharide consumption through the prebiotic product Bimuno.
  Interventions: Dietary Supplement: Bimuno Daily
- Placebo (Placebo Comparator): Maltodextrin powder
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bimuno Daily — Galactooligosaccharide supplement within Bimuno Daily
  Arms: GOS
Dietary Supplement: Placebo — Maltodextrin powder
  Arms: Placebo

SUMMARY:
Current evidence suggests that the amount of ingested carbohydrate that we can use for energy during exercise is limited by absorption levels in the gut. Thus, strategies to increase the amount of ingested carbohydrate our body can use are of great interest.

Recent evidence has shown we may be able to use more of the ingested carbohydrate during exercise when supplementing with probiotics ("good bacteria for our gut). It is currently unknown whether the food for these "good" bacteria (known as prebiotics) can induce a similar effect. Therefore, the purpose of this study is to understand if supplementation with the prebiotic Galactooligosaccharide (onwards referred to as BIMUNO®) can increase the use of ingested carbohydrate during exercise. We also aim to understand if BIMUNO® can enhance the availability of other nutrients, such as vitamins and minerals.

Participant will attend 8 laboratory sessions at the University of Bath. The first session is a screening visit lasting no more than 30 minutes. This can take place online, over the phone, or in-person, and the remaining 7 sessions will take place in a University of Bath laboratory. The next session is preliminary testing and familiarisation (approx. 2-2.5 hours). The remaining 6 visits (4 exercise trials & 2 baseline sample collection visits) will be split across 3 main blocks of the study, each lasting 28 days. Following preliminary testing, you will be randomised into supplementing with either BIMUNO®, or placebo. Block 1 will then begin with you attending the laboratory for a baseline sample collection visit, after which you will begin supplementation for the next 28 days. After this 28-day period, you will complete two exercise trials (details below). The ambient temperature in these trials (separated by >3 days) will differ (20 & 35˚C) and will occur in a random order. The second block (termed the 'washout' period) will be a 28-day period where you will take neither BIMUNO® nor the placebo. The third block will then commence and will be identical to block 1 - the only difference being you will take the alternative supplement.

ELIGIBILITY:
Inclusion Criteria:

* Regular exerciser - defined as participating in at least 30 mins of structured exercise at least 3 times per week
* Able to complete two hours of moderate intensity cycling
* Aged 18-60 years

Exclusion Criteria:

* Use of products marketed as prebiotics, probiotics or synbiotics within 4 weeks prior to study entry (e.g. Yakult, Actimel, Activia, VSL#3, Kefir). Regular cheese or yogurt containing lactic acid bacteria are not an exclusion criterion.
* Systemic antibiotic or antimycotic treatment within 4 weeks prior to study entry.
* Following diets likely to affect study outcomes: e.g. low FODMAP, KETO/high-fat, gluten free/coeliac, paleo, weight loss, caloric restriction, low-carb, 5:2/whole day energy restriction, Atkins/high-protein, sugar-free, single-food, juicing/any day of juicing, any other restriction diet (e.g. very low calory), or vegan diets (GOS is derived from cow's milk).
* Changes in diet, supplement use or medication likely to affect study outcomes within 2 months prior to study entry or planned during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Exogenous carbohydrate oxidation rate | 120 minutes
  amount of ingested carbohydrate used for energy within the body. measures in grams per minute and is calculated from breath samples

SECONDARY OUTCOMES:
Whole-body carbohydrate oxidation rate | 120 minutes
  measured from breath samples. unit is grams per minute
Whole-body fat oxidation rate | 120 minutes
  measured from breath samples. unit is grams per minute
Endogenous carbohydrate oxidation rate | 120 minutes
  measured from breath samples. unit is grams per minute
Blood lactate concentrations | 120 minutes
  measured from blood samples in millimoles per litre
Blood glucose concentrations | 120 minutes
  measured from blood samples in millimoles per litre
Plasma NEFA concentrations | 120 minutes
  measured from blood samples in micromoles per litre
Plasma insulin concentrations | 120 minutes
  measured from blood samples in picomoles per litre
Urinary calcium/creatinine ratio | 28 days
  measured from urine sample - ratio of milligrams per decilitre of calcium to milligrams per decilitre
Plasma 25-hydroxyvitamin D concentration | 28 days
  measured from blood samples. unit is nanomoles per litre
Plasma zinc concentration | 28 days
  measured from blood samples. unit is micrograms per decilitre
Plasma ferritin concentration | 28 days
  measured from blood samples. unit is micrograms per litre
Plasma vitamin B1 concentration | 28 days
  measured from blood samples. unit is micrograms per decilitre
Plasma vitamin B6 concentration | 28 days
  measured from blood samples. unit is micrograms per litre
Plasma vitamin C concentration | 28 days
  measured from blood samples. unit is micromoles per litre
Plasma vitamin E concentration | 28 days
  measured from blood samples. unit is micrograms per millilitre
Haemoglobin concentration | 120 minutes
  measured from blood samples. grams per decilitre
Haematocrit | 120 minutes
  measured from blood samples. unit is percentage of red blood cells in blood
Plasma intestinal fatty acid binding protein concentration | 120 minutes
  measured from blood samples. unit is nanograms per microlitre
Subjective scale: Gas | 120 minutes
  0-10 scale (0- no discomfort, 10- very severe discomfort)
Subjective scale: Regurgitation | 120 minutes
  0-10 scale (0- no discomfort, 10- very severe discomfort)
Subjective scale: Nausea | 120 minutes
  0-10 scale (0- no discomfort, 10- very severe discomfort)
Subjective scale: Fullness | 120 minutes
  0-10 scale (0- no discomfort, 10- very severe discomfort)
Subjective scale: Cramps | 120 minutes
  0-10 scale (0- no discomfort, 10- very severe discomfort)
Subjective scale: Urge to Defecate | 120 minutes
  0-10 scale (0- no discomfort, 10- very severe discomfort)
Rating of Perceived Exertion | 120 minutes
  Borg scale: 6-20. 6- very light, 20- extremely hard
Thermal Comfort | 120 minutes
  -4 to +4 scale. -4 very uncomfortable, 0 just comfortable, +4 very comfortable
Thermal Sensation | 120 minutes
  -4 to +4 scale. -4 very cold, 0 neutral, +4 very hot
Core temperature | 120 minutes
  measured via rectal probe
Skin temperature | 120 minutes
  measured via four temperature sensors. locations: chest, bicep, quadricep and gastrocnemius
Heart rate | 120 minutes
  measured via polar heart rate device placed on chest via strap

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Bath and NE Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No